CLINICAL TRIAL: NCT00205478
Title: A 12-Week, Double-Blind, Randomized, Parallel Group, Placebo Controlled Study of Two Doses of VX-702 in Subjects With Moderate to Severe Rheumatoid Arthritis
Brief Title: Phase 2 Clinical Study in Rheumatoid Arthritis With an Investigational Oral p38 MAP Kinase Inhibitor VX-702
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VX04-702-301
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — VX 702

INTERVENTIONS:
Drug: VX-702

SUMMARY:
The purpose of this study is to assess the clinical activity and safety of two doses of VX-702 compared to placebo in subjects with moderate to severe Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Adults with active rheumatoid arthritis for greater than 6 months and evidence of inflammation.

Exclusion Criteria:

* Subjects who have conditions precluding the use of cytokine inhibitors or subjects who require DMARDs other than hydroxychloroquine or sulfasalazine are excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-06; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for the study is the ACR20 response at Week 12.

SECONDARY OUTCOMES:
The ACR50 and ACR70 responses at 12 weeks will also be assessed as well as other measures.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kauffman, MD, PhD, Study Director — Vertex Pharmaceuticals Incorporated
Locations (43):
- Bulgaria (4):
  - Medical University - Sofia, Sofia
  - Military Medical Academy - Sofia, Sofia
  - Transport Hospital, Sofia
  - MBAL "Stara Zagora" EAD, Stara Zagora
- Croatia (3):
  - Thalassotherapia, Opatija
  - KBC Osijek Ambulanta za bol, Osijek
  - University Hospital Centre Zagreb, Zagreb
- Czechia (5):
  - University Hospital U Sv.Anny, Brno
  - Institute of Rheumatology, Prague
  - Rheumatology Out-patient Department, Prague
  - SZZ-Jizni Mesto II, Prague
  - University Hospital Kralovske Vinohrady, Prague
- Poland (9):
  - Szpital Specjalistyczny Nr 1, Bytom
  - Wojewodzki Szpital Zespolony, Elblag
  - Malopolskie Centrum Medyczne, Krakow
  - "Gabinety Profesorow" Prywatna Praktyka, Lublin
  - Instytut Medycyny Wsi im. Witolda Chodzki, Lublin
  - Wojewodzki Zespoￅﾂ Reumatologiczny im., Sopot
  - NZOZ "Nasz Lekarz" Praktyka Grupowa Lekarzy, Torun
  - Okregowy Szpital Kolejowy, Wroclaw
  - ZOZ Zyrardow, Żyrardów
- Russia (11):
  - Pirogov City Clinical Hospital #1, Moscow
  - State Institute of Rheumatology of RAMS, Moscow
  - State Clinical Immunology Research, Novosibirsk
  - Ryazan Regional Clinical Cardiologic, Ryazan
  - City Pokrovskaya Hospital, Saint Petersburg
  - EVIDENCE Clinical and Pharmaceutical Research, Saint Petersburg
  - Leningrad Regional Hospital, Saint Petersburg
  - Saint Petersburg Clinical Hospital, Saint Petersburg
  - Saint-Petersburg City Hospital, Saint Petersburg
  - Saint-Petersburg Medical Academy, Saint Petersburg
  - Saratov Regional Clinical Hospital, Saratov
- Serbia and Montenegro (3):
  - Institute of Rheumatology, Beograd
  - Institute of Rheumatology - Niska Banja, Niska Banja
  - Clinical Center Zemun, Zemun
- National Institute of Rheumatic Diseases, Piešťany, Slovakia
- Clinical Center Ljubljana, Ljubljana, Slovenia
- Ukraine (6):
  - Dniepropetrovsk State Medical Academy, Dniepropetrovsk
  - Donetsk State Medical University, Donetsk
  - Institute of Cardiology of Ukranian AMS, Kiev
  - Institute of Gerontology of Ukrainian AMS, Kiev
  - SanaClis s.r.o., Kiev
  - Zaporizhya Medical Institute, Zaporizhya

REFERENCES:
- [Derived] Damjanov N, Kauffman RS, Spencer-Green GT. Efficacy, pharmacodynamics, and safety of VX-702, a novel p38 MAPK inhibitor, in rheumatoid arthritis: results of two randomized, double-blind, placebo-controlled clinical studies. Arthritis Rheum. 2009 May;60(5):1232-41. doi: 10.1002/art.24485. PMID 19404957